CLINICAL TRIAL: NCT02174705
Title: A Randomized Controlled Trial of Rotavirus Vaccine vs. Sugar Water for Vaccine Injection Pain Management in Infants
Brief Title: Rotavirus vs. Sucrose for Vaccine Injection Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anna Taddio (Other)
Responsible Party: Sponsor-Investigator, Anna Taddio, Professor, University of Toronto
Organization: University of Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 30427
Record Dates: First submitted 2014-06-22; First posted 2014-06-25 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Vaccination Pain Management
Keywords: vaccination; pain management; sucrose; rotavirus
MeSH Terms: conditions — Agnosia | interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sucrose (Experimental): Sucrose prior to vaccine injections
  Interventions: Drug: Sucrose
- Rotavirus (Active Comparator): Rotavirus prior to vaccine injections
  Interventions: Drug: Rotavirus

INTERVENTIONS:
Drug: Sucrose — Sucrose 24% orally prior to vaccine injections
  Arms: Sucrose
Drug: Rotavirus — Rotavirus vaccine orally prior to vaccine injections
  Arms: Rotavirus

SUMMARY:
This randomized trial will compare the analgesic effectiveness of oral rotavirus vaccine to sugar water for reducing vaccine injection pain in infants.

ELIGIBILITY:
Inclusion Criteria:

* healthy infants receiving rotavirus vaccine in conjunction with primary immunizations in the first 6 months of life

Exclusion Criteria:

* impaired neurological development, history of seizures, sedatives or narcotics in preceding 24 hours, parent unable to use study tools, prior participation in the trial

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Distress | immediately after vaccinations in 15 seconds
  Observer rated using the Modified Behavioral Pain Scale (0-10) after each injection and overall

SECONDARY OUTCOMES:
Distress | immediately after vaccinations in 1 minute intervals for 2 minutes
  Observer rated cry duration after vaccination
Distress | immediately after vaccinations in 1 minute
  Immunizer rated distress after each injection using a Numerical Rating Scale (0-10)
Distress | immediately after vaccinations in 1 minute
  Parent rated distress after each injection using a Numerical Rating Scale (0-10)

OTHER OUTCOMES:
Safety | immediately after vaccinations in 5 minutes
  Number of infants spitting up/gagging with administration of study liquid
Satisfaction | immediately after vaccination in 1 minute
  Parent rated satisfaction with pain control using likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Anna Taddio, PhD, Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - Kindercare, Toronto, Ontario
  - Anna Taddio, Toronto, Ontario